CLINICAL TRIAL: NCT02988232
Title: Evaluation of the Efficacy and Safety of Herbal Medicine for Treating Work-related Chronic Low Back Pain: a Multicenter, Randomized, Controlled, Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Herbal Medicine for Treating Work-related Chronic Low Back Pain
Acronym: WRMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Sangji University Oriental Medical Center, Korea (Unknown); Semyung University Korean Medicine Hospital in Chungju, Korea (Unknown); Daejeon University (Other)
Responsible Party: Principal Investigator, Yun-Kyung Song, KMD PhD, Gachon University Gil Oriental Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISEE_2015_WRMD
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Low Back Pain; Workplace
Keywords: Work Related Chronic Low Back Pain; Korean Medicine; Sogyeonghwalhyeol-tang
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment(SGHH) (Experimental): Admission to Sogyeonghwalhyeol-tang granule
  Interventions: Drug: Sogyeonghwalhyeol-tang
- Placebo (Placebo Comparator): admission to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sogyeonghwalhyeol-tang — herbal extract
  Other Names: SGHH
  Arms: Treatment(SGHH)
Drug: Placebo — extract powder with same appearance, odor and color as SGHH
  Arms: Placebo

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of Sogyeonghwalhyeol-tang(SGHH) on Korean Patients With Work Related Chronic Low Back Pain

DETAILED DESCRIPTION:
Investigating the efficacy and safety of Sogyeonghwalhyeol-tang(SGHH) on Korean Patients With Work-related Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with chief complaint of low back pain in oriental rehabilitation medical center
* Age 19 - 65
* Workplace Vulnerable populations(hospital workers, office worker, blue collar workers, transit workers)
* Patients must include all of the following symptoms:

  * Those who have 4 ~7 cm of VAS pain score;
  * Those who has classified as 'at risk non-complier' or 'pain complaints' by KOSHA questionnaire
* Ability to have normal communication
* Ability to give informed consent

Exclusion Criteria:

1. Patients with pain duration of 3 months or less
2. Patients with progressive neurologic deficit or severe neurologic symptoms by SLR test
3. Patients diagnosed with serious pathology(s) which may cause low back pain (e.g. spinal metastasis of tumor(s), acute fracture, etc)
4. Patients with spondylolisthesis or spondylolysis(diagnosed with grade II or higher level)
5. Patients currently taking steroids, immunosuppressants, medicine for mental illness or other medication(s) that may interfere with study results
6. Patients with history of spinal surgery
7. Patients with more severe pain than pain caused by low back pain
8. Those who do not (cannot) abide by treatment and follow up due to the mental illness such as behavior disorder, depression, anxiety neurosis etc.
9. Patients with history of Medical Malpractice Case
10. Patients with treatment history of low back pain within 1 month either KM or WM
11. Patients participating in other clinical studies within 3 months
12. Pregnant patients or patients with plans of pregnancy or lactating patients
13. Patients disagree to sign the informed consent form
14. Patients deemed unsuitable for participating the trial by the researchers

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Numeric Rating Scale of Pain | Screening Visit, At baseline, week 2, 4, 6, 8
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) assesses the patients' current level of pain.

SECONDARY OUTCOMES:
Change from Baseline in 'Roland Morris Disability Questionnaire' | Screening Visit, At baseline, week 2, 4, 6, 8
  This is a self-reported questionnaire consisting of 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, bending over, sitting, lying down, dressing, sleeping, self-care and daily activities.
Change from Baseline in European Quality of life 5 Dimension | Screening Visit, At baseline, week 2, 4, 6, 8
  The EQ-5D is an international, standardized, generic instrument for describing and valuing health status. Participants were asked to indicate which of the following statements best describes their health state.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, PhD, Principal Investigator — Gachon University of Oriental Hospital
Locations (1):
- Gachon University Gil Oriental Medical Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided